CLINICAL TRIAL: NCT00558883
Title: Placebo Controlled Investigation on Action of Acarbose on the Sub-Clinical Inflammation and Immune Response in Early Type 2 Diabetes and Atherosclerosis Risk
Brief Title: AI(I)DA Acarbose and the Subclinical Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Technische Universität Dresden (Other); Diakonissen Krankenhaus Dresden, Germany (Unknown); University of Regensburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI(I)DA
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Type 2 Diabetes Mellitus; Subclinical Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): treatment with Acarbose: 2 weeks 1 x 50mg; 2 weeks 3 x 50mg; 16 weeks 3 x 100mg
  Interventions: Drug: acarbose
- 2 (Placebo Comparator): treatment with placebo: 2 weeks 1 x 50mg 2 weeks 3 x 50mg 16 weeks 3 x 100mg
  Interventions: Drug: acarbose

INTERVENTIONS:
Drug: acarbose — oral application

SUMMARY:
Acarbose an alphaglucosidase inhibitor changes in a complex way the transport, the digestion and the place of glucose release and absorption. As a result the intestinal milieu, the intestinal flora and the provision of enzymes in the lower small destine are changed. This should modify immune response of intestinal wall on food and its proinflammatory effects. The small intestine is the biggest immune organ of the organism. The postprandial glucose increase could have a direct effect on low-grade inflammation. Toxic effects (glucotoxicity), activation of the immune system and low grad inflammation could be reasons of developing endothelial dysfunction and affect plaque stability. The activity of the lymphocyte immune system in the intestine would be a further component, by which acarbose could take influence on diabetogenesis and atherogenesis. The question of an enterovasal axis is one of the new research concepts. As indicators of this axis considered: leucocytes, high sensitive C-reactive protein, plasminogen activator inhibitor antigen and lymphocytes sub-populations. The effect of acarbose on these parameters in the postprandial phase are not known yet.

DETAILED DESCRIPTION:
Acarbose, an alpha-glucosidase-inhibitor, delays the release of glucose out of complex carbohydrates in the upper small intestine. The digestion of carbohydrates after acarbose intake therefore mainly takes place in the lower small intestine and colon. Through this innovative mode of action the postprandial hyperglycemia is specifically delayed and flattened. Acarbose is used for more of 15 years for the therapy of type 2 diabetes. Efficiency and safety in treating diabetes were proved in extensive studies. Until today no serious side effects under acarbose were reported, the reduction of HbA1c is 0.7-1 %. Three large prospective studies and metaanalysis resp., could prove that acarbose has a highly significant positive effect on the incidence and progression of cardiovascular disease in people with prediabetes and type 2 diabetes resp. In the STOP-NIDDM-trail in persons with prediabetes as well as in the meta-analysis in type 2 diabetes (MERIA) the event rate in the acarbose group was ~ 50 % lower. In a substudy of the STOP-NIDDM intervention study a ca. 50 % lower progression of the intima-media-thickness of the A. carotis communis was documented under acarbose in comparison with placebo. In multivariate analysis acarbose was always the most important independent determinant of vasoprotective effects. Epidemiological investigations, even as controlled prospective studies, cannot establish causal relationships. Thus the question rises wether acarbose has - besides the known therapeutic effect on postprandial hyperglycemia pleiotropic effects, which lead to the documented preventive effects on cardiovascular complications. This would be of principal importance for the use of acarbose in patients with prediabetes / type 2 diabetes and increased vascular risk. So far acarbose is the only cardiovascular oral antidiabetic drug in people with IGT.

Working hypothesis:

Acarbose changes in a complex way the transport, the digestion and the place of glucose release and absorption. As a result the intestinal milieu, the intestinal flora and the provision of enzymes in the lower small intestine are changed. This should modify immune response of intestinal wall on food and its proinflammatory effects. The small intestine is the biggest immune organ of the organism. The postprandial glucose increase could have a direct effect on low-grade inflammation. Toxic effects (glucotoxicity), activation of the immune system and low-grade inflammation could be reasons of developing endothelial dysfunction and affect plaque stability. The activity of the lymphocyte immune system in the intestine would be a further component, by which acarbose could take influence on diabetogenesis and atherogenesis. The question after an enterovasal axis is now one of the most fascinating new research concepts and basis of incretin-related drug treatment of diabetes resp. As intravasal indicator for low-grade inflammation are considered: leucocytes, high sensitive C-reactive protein (hsCRP) and plasminogen activator inhibitor active antigen (PAI1) as well as lymphocytes subpopulations. The effects of acarbose on these parameters in the postprandial phase are not known yet.

ELIGIBILITY:
Inclusion criteria:

In this study patients with type 2 diabetes are included, who fulfil the following criteria:

* type 2 diabetes by WHO criteria, aged 30-75
* HbA1c ≥ 6.5 % < 8.0 % and/or 2h 75 OGTT plasma glucose ≥ 11.1 mmol/l
* fasting leucocytes count ≥ 6.2 GPt/l (median for newly diagnosed type 2 patients in RIAD) and/or hsCRP ≥ 1.0 mg/dl and < 10 mg/dl (earlier 2.8 mg/dl)
* informed consent

Exclusion criteria:

Excluded were patients with one of the following criteria:

* contraindication for acarbose
* chronic gastrointestinal disease
* prior antidiabetic treatment
* intake of statins or drugs with antiinflammatory effects
* acute or chronic inflammatory diseases
* MI or stroke < 6 months before entry
* immune diseases
* neoplasia
* diseases with acute weight loss

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
effect of treatment of leucocyte count before and after test meal | 20 weeks

SECONDARY OUTCOMES:
identification of gene arrays are registered of relevant pharmacodynamic structures and metabolism ways. Histological examinations of bioptats; Blood: hsCRP, PAI1; Lymphocyte subpopulations; blood lipids, plasma glucose fasting and postprandial | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Markolf Hanefeld, PhD, MD, Principal Investigator — GWT-TUD GmbH, Centre for Clinical Studies
Locations (1):
- GWT-TUD GmbH; Centre for Clinical Studies, Dresden, Germany